CLINICAL TRIAL: NCT02287961
Title: Natural History of Anal Human Papillomavirus Infection and Associated Disease in HIV-infected Men Who Have Sex With Men: Towards an Evidence Base for the Prevention of Anal Cancer.
Brief Title: Human Papillomavirus Infection and Related Anal Lesions in HIV-positive Men Who Have Sex With Men
Acronym: APACHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS EP57 APACHES
Record Dates: First submitted 2014-10-15; First posted 2014-11-11 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hiv Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects (Other): * Standard proctologic examination with digital rectal examination and 2 anal swabs at initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits
  * High resolution anoscopy at initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits
  * Biopsy(ies) during High Resolution Anoscopy only if lesion suggestive of AIN detected during High Resolution Anoscopy
  * High Resolution Anoscopy biannually only if high-grade lesion (ASC-H, HSIL ou AIN2/3)
  Interventions: Procedure: Standard proctologic examination; Procedure: High resolution anoscopy; Procedure: Biopsy(ies) during High Resolution Anoscopy; Procedure: High Resolution Anoscopy biannually

INTERVENTIONS:
Procedure: Standard proctologic examination — (with digital rectal examination and 2 anal swabs) at initial inclusion visit, M12 and M24 follow-up visits and if applicable M6 and M18 control visits
Procedure: High resolution anoscopy — at initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits
Procedure: Biopsy(ies) during High Resolution Anoscopy — only if lesion suggestive of AIN detected during High Resolution Anoscopy
Procedure: High Resolution Anoscopy biannually — Only if high-grade lesion (ASC-H, HSIL ou AIN2/3)

SUMMARY:
Multicentric epidemiological non-comparative study in France characterising evolution of anal Human papillomavirus (HPV) infection and related lesions and evaluating markers associated with the observed evolution.

Estimated enrolment: 500

Principal Outcomes

* Detection of high-grade cytological and histological anal lesions by high resolution anoscopy
* Spontaneous regression of high-grade anal lesions
* Detection of anal HPV infection

Intervention (procedure):

* Patient medical interview (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)
* Standard proctologic examination with digital rectal examination and 2 anal swabs (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)
* High resolution anoscopy (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)

Only if lesion suggestive of Anal Intraepithelial Neoplasia (AIN) detected during High Resolution Anoscopy (HRA):

- anal biopsy(ies) during HRA

Only if high-grade lesion:

- HRA biannually

DETAILED DESCRIPTION:
Intervention (procedure):

* Patient medical interview (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)
* Standard proctologic examination with digital rectal examination and 2 anal swabs (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)
* High resolution anoscopy (initial inclusion visit, Month 12 and Month 24 follow-up visits and if applicable Month 6 and Month 18 control visits)

Only if lesion suggestive of Anal Intraepithelial Neoplasia (AIN) detected during High Resolution Anoscopy (HRA):

- anal biopsy(ies) during HRA

Only if high-grade lesion (Atypical squamous cells-cannot exclude high-grade squamous intraepithelial lesion (ASC-H), High grade Superficial Intra-epithelial Lesion (HSIL) or AIN2/3):

- HRA biannually

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* At least 35 years old
* HIV-positive (documented search of HIV infection, with HIV status determined according to HAS algorithm)
* Signed informed consent
* Affiliated to or beneficiary of French social security
* All severity criteria and evolution of HIV disease are accepted (including AIDS stage and co-infections)

Exclusion Criteria:

* Contraindication to biopsy
* History of anal cancer or pelvic radiotherapy
* AIN2/3 treated during previous year
* Current anticancer chemotherapy or within 24 months before inclusion
* Difficulty in evaluation (anus reshaped and/or scarred)
* Individual placed under judicial protection
* Foreseen absence which may hamper participation; insufficient motivation; associated pathology with priority for care

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of high-grade anal lesions by high resolution anoscopy | Initial inclusion visit
Evaluation of anal HPV infection by DNA, RNA and protein detection | Initial inclusion visit
Quantification of spontaneous regression of high-grade anal lesions | Month 24

SECONDARY OUTCOMES:
Evaluation of anal HPV infection by DNA, RNA and protein detection | Month 6
Evaluation of anal HPV infection by DNA, RNA and protein detection | Month 12
Evaluation of anal HPV infection by DNA, RNA and protein detection | Month 18
Evaluation of anal HPV infection by DNA, RNA and protein detection | Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Etienney, Principal Investigator — Hôpital Diaconesses Paris; Gary Clifford, Study Director — International Agency for Research on Cancer
Locations (1):
- Diaconesses, Paris, France

REFERENCES:
- See also: Agence nationale de recherches sur le sida et les hépatites virales (ANRS) — http://anrs.fr